CLINICAL TRIAL: NCT01254123
Title: Effect of Additional Treatment With EXenatide in Patients With an Acute Myocardial Infarction (the EXAMI Trial)
Acronym: EXAMI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL28593.029.09
Record Dates: First submitted 2010-11-29; First posted 2010-12-06 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2010-01

CONDITIONS: Patients With a First Acute Myocardial Infarction to be Treated With Primary Percutaneous Coronary Intervention (PCI).
Keywords: Glucagon Like Peptide-1; Exenatide; myocardial infarction; MRI; PCI
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide (Active Comparator)
  Interventions: Drug: Exenatide infusion
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo infusion.

INTERVENTIONS:
Drug: Exenatide infusion — On arrival to our cardiac care unit (CCU) and after informed consent patients will be randomized to Exenatide infusion or Placebo infusion. Patients in the Exenatide group will immediately be treated be with Exenatide iv, 5ug bolus in 30 minutes, followed by a continuous Exenatide infusion of 20ug/ 24 hours.
  Exenatide preparation: Byetta injection pens containing 1,2 ml (concentration 0,25 mg/ml; 60 doses of 5 μg) will be obtained. 3 doses (15 μg) will be diluted in 49 ml saline and 1 ml Human Serum Albumen (Cealb 200g/L, 10ml) to get a total of 50 ml containing 15 μg exenatide (or 300 ng exenatide / ml). A 50cc syringe will be placed in a pump system that is connected with a cannula in the patient's vein. The infusionrate will be 33,3 ml/hr for the first 30 minutes, followed by an infusion rate of 2,8 ml/hr for 72 hours. New 50cc syringes will be made every 8 hours.
  Arms: Exenatide
Drug: Placebo infusion. — On arrival to our cardiac care unit (CCU) and after informed consent patients will be randomized to Exenatide infusion or Placebo infusion. Patients in the placebo group will immediately be treated with placebo infusion.
  Placebo preparation: 49ml saline and 1ml Human Serum Albumen (Cealb 200g/L, 10ml) to get a total of 50 ml will be placed in a 50cc syringe and placed in a pump system that is connected with a cannula in the patient's vein. The infusionrate will be 33,3 ml/hr for the first 30 minutes, followed by an infusion rate of 2,8 ml/hr for 72 hours. New 50cc syringes will be made every 8 hours.
  Arms: Placebo

SUMMARY:
Myocardial infarction (MI) causes loss of myocytes and may lead to loss of ventricular function, morbidity and mortality. The most effective therapy is early reperfusion of the ischemic myocardium by percutaneous coronary intervention (PCI). Reperfusion limits myocardial ischaemic necrosis, but also induces inflammation, oxidative stress and calcium overload: a process referred to as reperfusion injury leading to necrosis and apotosis. Glucagon Like Peptide-1 (GLP-1) is an incretin hormone that has shown to activate anti-apoptotic enzymes, reducing reperfusion injury. GLP-1 agonists have been demonstrated to be cardioprotective in several animal studies and in a single small non-randomized clinical study. In this pilot study we will assess the safety and efficacy of GLP-1 receptor agonist Exenatide infusion compared to placebo in patients with an acute myocardial infarction undergoing primary PCI.

A total of 40 patients will be included in this single centre prospective randomised placebo controlled two-arm pilot study. Patients who are to undergo a primary PCI for a first acute ST elevation myocardial infarction are randomly assigned to placebo or Exenatide 5ug bolus in 30 minutes, followed by a continuous Exenatide infusion of 20ug/ 24 hours for 72 hours. Blood samples are obtained for assessment of enzymatic infarct size and Exenatide levels. Side effects of Exenatide are stringently monitored. Cardiac function will be measured using Cardiac Magnetic Resonance Imaging (CMRI) and 3D echocardiography at 1 week and 4 months post MI. Infarct size will be assessed by means of the final infarct size at 4 months post MI as a percentage of the area at risk at 1 week post MI. Furthermore we will compare the RNA profile of both groups.

ELIGIBILITY:
Inclusion Criteria:

* >18 and < 80 years of age
* First myocardial infarction
* ST elevation of more than one mm in at least 2 separate leads on the electrocardiogram (ECG)
* Delay between onset of sustained chestpain and PCI < 6 hours.

Exclusion Criteria:

* Cardiac rhythm is other than normal sinus rhythm.
* Patient in Killip class 3 or 4 of heart failure
* Cardiogenic shock defined as sustained systolic blood pressure ≤ 80mmHg despite fluid hydration.
* Post cardiac resuscitation
* Need for intra aortic balloon counterpulsation therapy
* The patient is unable to hold his/her breath for up to 20 seconds due to age or concomitant illness
* No former PCI performed
* No recanalisation achieved of the occluded coronary artery
* Culprit not in segment 1,2,3,6,7,11,12,13 of the coronary artery
* No definite culprit
* More than one occluded vessel, or a more than 70% stenosis by visual assessment in a non-culprit vessel.
* TIMI 3 flow in culprit lesion at presentation
* Decreased renal function eGFR < 30ml/min
* Any contraindication for MRI ie: implanted electronic devices such as pacemakers, internal defibrillators, neurostimulators, implanted drug infusion devices, cochlear implants, cerebrovascular clips, claustrophobia. previous vascular surgery: aneurysm clip, carotid artery vascular clamp, aortic clips, venous umbrella spinal/intra-ventricular shunts
* Metal fragments in eye, head, ear, skin or shoulder.
* Swann-Ganz catheter.
* Known pre-existing left ventricular dysfunction measured by any technique (ejection fraction < 45% prior to current admission for myocardial infarction)
* Prior myocardial infarction
* Prior coronary artery bypass grafting
* Moderate to severe cardiac valve disease
* Stroke or transient ischemic attack within the previous 24 hours
* Serious known concomitant disease with a life expectancy of less than one year
* Follow up impossible
* Previous participation in a trial within the previous 30 days
* Known type I Diabetes Mellitus
* Known type II Diabetes Mellitus
* Pregnancy and/or lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-11

PRIMARY OUTCOMES:
Safety of GLP-1 receptor agonist Exenatide infusion compared to placebo in patients with an acute myocardial infarction undergoing primary PCI

SECONDARY OUTCOMES:
Infarct size, assessed by means of the final infarct size at 4 months post myocardial infarction (CMRI) as a percentage of the area at risk at 1 week post myocardial infarction (T2 weighed CMRI).
Regional myocardial function based on a MRI segmental analysis at 1 weeek and at 4 months post myocardial infarction.
Global left ventricular ejection fraction (EF), Left Ventricular End Systolic Volume (LVESV), Left Ventricular End Diastolic Volume (LVEDV) at 1 week and at 4 months post myocardial infarction measured by Cardiac MRI.
Regional myocardial function assessed by 2D and 3D echocardiography at 1 week and at 4 months post myocardial infarction.
Global left ventricular EF, LVESV, LVEDV at 1 week and at 4 months post myocardial infarction measured by 2D and 3D echocardiography.
Angiographic parameters as Trombolysis In Myocardial Infarction (TIMI) frame count and TIMI blush grade after PCI.
The occurrence within 4 months of a Major Adverse Cardiac Event (MACE) defined as cardiac death, myocardial infarction, coronary bypass grafting, or a repeat PCI .
Side effects of exenatide
Serum-glucose levels during the first 72 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Yolande Appelman, Dr., Principal Investigator — Dept. of Cardiology VU Medical Center
Locations (1):
- VU Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Huang M, Wei R, Wang Y, Su T, Li Q, Yang X, Chen X. Protective effect of glucagon-like peptide-1 agents on reperfusion injury for acute myocardial infarction: a meta-analysis of randomized controlled trials. Ann Med. 2017 Nov;49(7):552-561. doi: 10.1080/07853890.2017.1306653. Epub 2017 Mar 31. PMID 28286967
- [Derived] Scholte M, Timmers L, Bernink FJ, Denham RN, Beek AM, Kamp O, Diamant M, Horrevoets AJ, Niessen HW, Chen WJ, van Rossum AC, van Royen N, Doevendans PA, Appelman Y. Effect of additional treatment with EXenatide in patients with an Acute Myocardial Infarction (EXAMI): study protocol for a randomized controlled trial. Trials. 2011 Nov 8;12:240. doi: 10.1186/1745-6215-12-240. PMID 22067476